CLINICAL TRIAL: NCT07320859
Title: Mirror Therapy Versus Music Therapy for Pain During Arteriovenous Fistula Cannulation in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Comparing Mirror and Music for Dialysis Needle Pain
Acronym: MIRROR-MUSIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Kavram Vocational School (Other)
Collaborators: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Izmir Kavram, Assistant Professor Dr, Izmir Kavram Vocational School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22.10.2025/2544
Record Dates: First submitted 2025-12-15; First posted 2026-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Pain, Procedural; Arteriovenous Fistula
Keywords: Mirror Therapy; Music Therapy; Non-pharmacological Pain Management; Hemodialysis; Vascular Access; Cannulation Pain
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pain, Procedural; Arteriovenous Fistula | interventions — Mirror Movement Therapy; Music Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1:1 ratio to one of three parallel groups for the duration of the study.
Masking Description: Due to the nature of the interventions (music listening and mirror viewing), participants and the nurses providing care were not blinded to group assignment. However, the statistician who performed the final data analysis was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror group (Experimental): During arteriovenous fistula cannulation, patients viewed the reflection of their healthy arm in a 40-cm mirror placed approximately 30 cm away. They focused on this image for 10 minutes before cannulation (adaptation phase), and the procedure was performed while they continued to look at the mirror. The visual illusion aimed to modulate pain perception.
  Interventions: Device: Mirror Therapy (Visual Illusion Therapy)
- Music group (Experimental): During arteriovenous fistula cannulation, patients listened to pre-selected, calming instrumental Turkish classical music (Nihavend and Muhayyerkürdi maqams) via headphones and an MP3 player at a comfortable volume. The music started before cannulation and continued throughout the procedure.
  Interventions: Other: Music Therapy
- Control group (No Intervention): Patients received routine, standard cannulation care as per the hemodialysis unit protocol, without any additional non-pharmacological intervention such as mirror or music therapy.

INTERVENTIONS:
Device: Mirror Therapy (Visual Illusion Therapy) — A non-pharmacological, behavioral intervention. A standard mirror (40 cm diameter) is positioned to allow the patient to view the reflection of their non-cannulated, healthy arm during arteriovenous fistula cannulation. The patient focuses on this visual illusion for an adaptation period (10 minutes) before the needle insertion. The intervention is based on the principles of graded motor imagery and aims to reduce procedural pain by modulating cortical representation and attention.
  Arms: Mirror group
Other: Music Therapy — A non-pharmacological, complementary therapy. Patients listen to pre-recorded, instrumental Turkish classical music (specifically Nihavend and Muhayyerkürdi maqams) via headphones during the cannulation procedure. The music is selected for its calming properties and starts before needle insertion. The intervention aims to reduce pain and anxiety through auditory distraction, emotional modulation, and relaxation.
  Arms: Music group

SUMMARY:
Inserting needles into the vascular access (fistula) is a major source of pain and anxiety for many hemodialysis patients. This study compared two simple, non-drug techniques to reduce this pain: listening to music and looking into a mirror during the needle insertion.

A total of 75 adult patients receiving regular hemodialysis at Izmir Özel Can Dialysis Center were randomly divided into three groups: a music group, a mirror group, and a control group. Patients in the music group listened to calming, instrumental Turkish classical music (makam) via headphones during cannulation. Patients in the mirror group looked at the reflection of their healthy arm in a mirror. The control group received standard care without these interventions.

Pain intensity was measured immediately after needle insertion using a 10-cm Visual Analogue Scale (VAS), where 0 means "no pain" and 10 means "the worst imaginable pain." Pain scores were compared between the groups to determine which method was more effective.

The results of this study may provide nurses and patients with easy-to-use, evidence-based options to make hemodialysis needle procedures less painful and stressful.

DETAILED DESCRIPTION:
Study Design: This was a prospective, three-arm, parallel-group, randomized controlled trial with a 1:1:1 allocation ratio.

Setting and Sample: The study was conducted at the Hemodialysis Unit of Izmir Özel Can Dialysis Center between December 1 and 30, 2025. The study population consisted of 150 patients. The sample size was calculated using G*Power 3.1.9.2 software. With a significance level (alpha) of 0.05, a power (1-beta) of 80%, and an effect size of 5%, a sample of 25 patients per group (total n=75) was determined to be sufficient for a three-group comparison.

Inclusion Criteria:

Age between 18 and 85 years.

Receiving hemodialysis treatment three times per week.

Literate (able to read and write).

No hearing impairment.

Native Turkish speaker.

On hemodialysis for at least 6 months.

Baseline pain score >3 on the Visual Analogue Scale (VAS).

Willing to listen to music.

Exclusion Criteria:

Presence of a psychological disorder.

Communication problems.

Diagnosis of cancer.

Unwillingness to participate in the study.

Randomization: Eligible patients were randomly assigned to one of three groups: the Music Intervention Group, the Mirror Intervention Group, or the Control Group.

Interventions:

Music Intervention Group: During the arteriovenous fistula (AVF) cannulation procedure, patients listened to pre-selected instrumental Turkish classical music (makam), specifically Nihavend and Muhayyerkürdi maqams, via an MP3 player and headphones. The volume was adjusted to a comfortable level.

Mirror Intervention Group: During cannulation, a standard mirror (40 cm in diameter) was positioned on a table stand. It was adjusted so that patients could see the reflection of their healthy (non-cannulated) arm. The distance between the fingertips of the reflected hand and the mirror surface was approximately 30 cm. Patients were instructed to focus only on the image of their healthy hand in the mirror. The cannulation was performed in two phases: immediately after looking at the healthy hand image (incongruent phase) and after 10 minutes of adaptation to the mirror image (adaptation phase).

Control Group: Patients received standard cannulation care without any additional intervention.

Data Collection Tools:

Patient Information Form: Collected socio-demographic characteristics, dialysis duration, and details about pain (location, intensity, type, timing, cause, and coping methods).

Visual Analogue Scale (VAS): A 10-cm horizontal line used to measure pain intensity, where the left end (0 cm) represents "no pain" and the right end (10 cm) represents "the worst pain imaginable." Patients marked their current pain level on the line, and the distance from the left end was measured in centimeters to obtain a numerical score (0-10).

Procedure: After providing informed consent, all participants completed baseline assessments (Patient Information Form, VAS). The interventions were applied during subsequent cannulation sessions as described. Procedural pain was assessed using the VAS immediately after cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-85 years of age or older

  * Receiving HD treatment 3 days a week
  * Being able to read and write
  * Having no hearing impairment
  * Having Turkish as their native language
  * Having received HD treatment for at least 6 months
  * Having a VAS pain score >3
  * Agreeing to listen to music

Exclusion Criteria:

* Having a psychological disorder

  * Having communication problems
  * Having cancer
  * Not wanting to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Procedural pain intensity during arteriovenous fistula cannulation | Procedure (during cannulation)
  Pain intensity experienced by the patient immediately following the needle insertion for hemodialysis. This primary outcome is measured during the second and third hemodialysis sessions following randomization (the first session post-randomization served as a runin with no intervention). Pain is measured using a 10-cm Visual Analogue Scale (VAS). Scores range from 0 to 10, where 0 cm represents 'no pain' and 10 cm represents 'the worst pain imaginable,' and higher scores indicate worse pain (greater pain intensity). The patient marks their pain level on the line, and the score is recorded in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Kavram Vocational School, Konak, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated during this study are not publicly available due to the small sample size and the potential risk of compromising individual privacy, even after de-identification. However, anonymized data may be made available from the corresponding author upon reasonable request and with permission from the institutional ethics committee.